CLINICAL TRIAL: NCT00733187
Title: A Pharmacokinetic Study to Evaluate the Effect of Food on the Oral Bioavailability and Effect of Diurnal Variation on the Pharmacokinetics of ABT-869
Brief Title: Pharmacokinetic Study To Evaluate Effect of Food and Diurnal Variation on ABT-869
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M10-384
Record Dates: First submitted 2008-08-08; First posted 2008-08-12 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2013-01

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: ABT-869

INTERVENTIONS:
Drug: ABT-869 — 0.25 mg/kg

SUMMARY:
To estimate the effect of food on the oral bioavailability and effect of diurnal variation on the pharmacokinetics of ABT-869.

DETAILED DESCRIPTION:
This study is a pharmacokinetic study designed to evaluate the effect of food on the oral bioavailability and effect of diurnal variation on the pharmacokinetics of ABT-869. Triplicate ECG performed to determine the effect of ABT-869 on QT prolongation . Subjects may continue receiving linifanib after completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age is ≥ 18 years.
* Must have a histologically or cytologically confirmed non-hematologic malignancy that is refractory to standard therapies or for which a standard effective therapy does not exist.
* Has measurable or evaluable disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0-2.
* Must have adequate bone marrow, renal and hepatic function as follows:

  * Bone Marrow: Absolute neutrophil count (ANC) ≥ 1,500/mm³; Platelets ≥ 100,000/mm³; Hemoglobin ≥ 9.0 g/dL (1.4 mmol/L)
  * Renal function: serum creatinine ≤ 2.0 mg/dL (0.81 mmol/L);
  * Hepatic function: AST and ALT ≤ 1.5 × ULN unless liver metastases are present, then AST and ALT ≤ 5.0 × ULN; bilirubin ≤ 1.5 mg/dL (0.026 mmol/L)
* Must have PTT ≤ 1.5 × ULN and/or INR ≤ 1.5 .
* Women of childbearing potential and men must agree to use adequate contraception (one of the following listed below) prior to study entry, for the duration of study participation and up to two months following completion of therapy. Women of childbearing potential must have a negative urine pregnancy test within 7 days prior to initiation of treatment and/or post menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.

  * total abstinence from sexual intercourse (minimum one complete menstrual cycle);
  * a vasectomized partner;
  * hormonal contraceptives (oral, parenteral or transdermal) for at least 3 months prior to study drug administration;
  * intrauterine device; * double-barrier method (condoms, contraceptive sponge, diaphragm or vaginal ring with spermicidal jellies or cream)
* Is capable of understanding and complying with parameters as outlined in the protocol and able to sign the informed consent.
* Must voluntarily sign and date each informed consent, approved by an Independent Ethics Committee (IEC)/Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* Has received anti-cancer therapy within 21 days or within a period defined by 5 half lives, whichever is shorter, prior to study drug administration. Has not recovered to less than or equal to Grade 1 clinically significant adverse effects/toxicities of the previous therapy. Avastin must not have been used less than 60 days prior to receiving ABT-869.
* Has had major surgery within 21 days of Study Day 1.
* Has untreated brain or meningeal metastases. Subjects with treated, stable, asymptomatic central nervous system lesions may be considered. Subject must have had stable disease for at least 4 weeks prior to study entry.
* Has been diagnosed with hepatocellular carcinoma.
* Pregnant or breastfeeding female.
* Is receiving therapeutic anticoagulation therapy. Low dose anticoagulation for catheter prophylaxis will be permitted.
* Has a history of/or currently exhibits clinically significant cancer related events of bleeding. The subject has a recent history of (within 4 weeks of Study Day 1) or currently exhibits other clinically significant signs of bleeding.
* Has proteinuria CTC Grade > 1 at baseline as measured by a UPC ratio of > 1 and confirmed by a 24 hour urine collection. . Currently exhibits symptomatic or persistent, uncontrolled hypertension defined as diastolic blood pressure (BP) > 100 mmHg; or systolic blood pressure (BP) > 150 mmHg.
* Has a history of myocardial infarction within 6 months of Study Day 1.
* Has known autoimmune disease with renal involvement.
* Is receiving combination anti-retroviral therapy for human immunodeficiency virus (HIV).
* Clinically significant uncontrolled condition(s).
* Has active ulcerative colitis, Crohn's disease or celiac disease.
* LV Ejection Fraction < 50%.
* Current or previous enrollment in another clinical study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic | Various timepoints
  Blood samples for the pharmacokinetics of linifanib will be collected for each subject and each regimen (fasting, fed, AM and PM dosings).
ECG Evaluation | Various timepoints
  Triplicate ECG will be performed at designated timepoints.
Adverse Events | Throught the study
  Only treatment emergent AEs will be included. Toxicity grade, relationship to study drug and AEs leading to discontinuation will be evaluated.
Lab data and vital signs | Various timepoints
  Blood chemistry and hematology will be analyzed based on the regimen and dosing and overall. 24 hr ABPM will be analyzed by regimen and dosing time and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Ricker, MD, Study Director — AbbVie

REFERENCES:
- [Result] Xiong H, Chiu YL, Ricker JL, LoRusso P. Results of a phase 1, randomized study evaluating the effects of food and diurnal variation on the pharmacokinetics of linifanib. Cancer Chemother Pharmacol. 2014 Jul;74(1):55-61. doi: 10.1007/s00280-014-2475-z. Epub 2014 May 9. PMID 24810181
- [Derived] Chiu YL, Lorusso P, Hosmane B, Ricker JL, Awni W, Carlson DM. Results of a phase I, open-label, randomized, crossover study evaluating the effects of linifanib on QTc intervals in patients with solid tumors. Cancer Chemother Pharmacol. 2014 Jan;73(1):213-7. doi: 10.1007/s00280-013-2351-2. Epub 2013 Nov 16. PMID 24241212